CLINICAL TRIAL: NCT03140384
Title: Compare the Different Routes of Administration of Misoprostol During Medicinal Abortion Between 7 and 9 Weeks of Amenorrhoea (SA)
Acronym: Misoprostol
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no regulatory approval
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016_843_0033
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Misoprostol; Drug-induced Abortion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Administration of oral Misoprostol (Active Comparator)
  Interventions: Biological: Assess the efficacy and side effects of Misoprostol according to the route of administration
- Administration of Misoprostol vaginally (Active Comparator)
  Interventions: Biological: Assess the efficacy and side effects of Misoprostol according to the route of administration
- Administration of buccal Misoprostol (Active Comparator)
  Interventions: Biological: Assess the efficacy and side effects of Misoprostol according to the route of administration

INTERVENTIONS:
Biological: Assess the efficacy and side effects of Misoprostol according to the route of administration — Assess the efficacy and side effects of Misoprostol according to the route of administration

SUMMARY:
In France, drug-induced abortion is allowed up to 9SA, after which the surgical route is preferred. Mifepristone 600mg is used 36-48 hours before the introduction of Misoprostol. This is recommended orally at a dose of 400 μg. There are currently several studies on the subject, including a meta-analysis of the 2011 Cochrane Database, but doses, routes of administration and gestational age differ in all studies. Currently, HAS recommends the vaginal route at the dose of 800μg for stopped pregnancies. It is therefore necessary to compare the different routes of administration of Misoprostol at the same dose to allow to change our French recommendations on the medicinal abortion and perhaps also to recommend the vaginal route in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years hospitalized using abortions between 7 and 9 SA and after informed consent,
* Affiliation to a social security scheme.

Exclusion Criteria:

* Minor or major women under guardianship or curatorship
* BMI <18.5 (thinness)
* Ambulatory
* Several abortions on the duration of the study
* Take Mifepristone> 48 hours before taking Misoprostol
* Contraindications to Misoprostol: Prostaglandin Allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2019-07-20 (Estimated); Study Completion 2019-07-20 (Estimated)

PRIMARY OUTCOMES:
Complete pregnancy evacuation on ultrasound at 3 weeks | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France